CLINICAL TRIAL: NCT00241176
Title: Open Label Trial of Aripiprazole in Children and Adolescents With Tourette's Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H12189
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Results first posted 2013-01-25 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-10

CONDITIONS: Tourette's Syndrome; Tic Disorders
Keywords: Psychiatric; Clinical Trial; Pediatrics; Tourette's Disorder; Tic Disorder
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aripiprazole (Experimental)
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Baseline Visit 2: Subjects btw 25-50kg start on 1.25mg/day, btw 50-70kg start on 2.5mg/day, greater than 70kg start on 5mg/day Visit 3: Titrated based on YGTSS & CGI-TS ratings at investigator discretion. Subjects who show evidence of response (reduction in CGI-TS by 1-2 points) may remain on same dose. Subjects who show no response may increase as follows: btw 25-50kg increase to 2.5mg/day, btw 50-70kg increase to 3.75mg/day, greater than 70kg increase to 7.5mg/day Visit 5: Subjects who show no response may increase as follows: btw 25-50kg increase to 3.75mg/day, btw 50-70kg increase to 5mg/day, greater than 70kg increase to 10mg/day Visit 6: Subjects who show no response may be increase as follows: btw 25-50kg increase to 5mg/day, btw 50-70kg increase to 7.5mg/day, greater than 70kg increase to 12.5mg/day Visit 7: Subjects who how no response may be increase as follows: btw 25-50kg increase to 7.5mg/day, btw 50-70kg increase to 10mg/day, greater than 70kg increase to 15mg/day

SUMMARY:
The purpose of this study is to determine if Abilify will reduce tics (repetitive, uncontrollable movements or vocalizations) in children and adolescents ages 7-18 with Tourette's Disorder (TD) or a chronic motor tic disorder (either repetitive, uncontrollable movements or vocalizations).

DETAILED DESCRIPTION:
The aims of this study are to obtain systematic data regarding dosing and safety of aripiprazole (Abilify) in the treatment of youth with Tourette's Disorder (TD). Tourette's Disorder is characterized by multiple motor (more than one uncontrollable movement) and vocal tics (vocal outbursts) which have been present for more than 1 year, with onset before the age of 18. The disorder causes marked distress in social, occupational or other important areas of functioning. Abilify has been approved by the United States Food and Drug Administration (FDA) to treat adults with schizophrenia but has not been approved to treat Tourette's Disorder (TD) so it is considered experimental or investigational in this study.

ELIGIBILITY:
Inclusion Criteria:

* Child or adolescent must be 7 to 18 years of age (inclusive) when informed consent is obtained.
* Must meet full criteria for Tourette's Disorder or chronic motor tic disorder.
* Must have failed to respond to an adequate trial, as determined by the investigator, of clonidine, guanfacine, or neuroleptic medication in the past.
* Tics are causing significant distress or impairment, as determined by parent/subject and principal investigator, on current treatment regimen.
* Laboratory results, including serum chemistries, hematology, and urinalysis, must show no significant abnormalities (significant is defined as laboratory values requiring acute medical intervention).
* Must be able to swallow pills.
* Must be of normal intelligence in the judgment of the investigator.
* Must possess an educational level, degree of understanding and command of the English language to enable them to communicate suitably with the investigator and study coordinator, and to understand the nature of the study.
* Subjects and their legal representatives must be considered reliable.
* Written informed consent of parents and subjects (ages 18 and above) and assent of subjects ages 7-17 will be obtained.

Exclusion Criteria:

* Organic brain disease, for example, traumatic brain injury residua.
* Mental retardation as defined by the DSM-IV-TR.
* A history of seizure disorder (other than febrile seizure).
* A history of Sydenham's Chorea.
* Autism, schizophrenia, other psychotic disorder, or bipolar disorder.
* A primary diagnosis of a major mood disorder that requires ongoing psychiatric treatment.
* A neurological disorder other than a tic disorder.
* A major medical illness.
* Females who are of child bearing age who are unwilling to use birth control or who are pregnant, as determined by serum pregnancy test at baseline assessment, or lactating.
* Have a past or current history of substance dependence and/or a current history of substance abuse or who fail baseline toxic screen.
* Have any clinically significant abnormal laboratory result at baseline screening including EKG, or blood tests.
* Have a history of ongoing or previously undisclosed child abuse (risk of removal from home would not allow for consistent caretaker ratings).

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2005-09; Primary Completion 2008-08 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Coffey, M.D, M.S., Principal Investigator — NYU School of Medicine, NYU Child Study Center
Locations (1):
- NYU Child Study Center, New York, New York, United States

REFERENCES:
- See also: NYU Child Study Center website — http://www.aboutourkids.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Aripiprazole: Subjects received initial dose based on body weight at Visit 2: Subjects between 25-50 kg were started on 1.25 mg/day, Subjects between 50-70 kg were started on 2.5 mg/day, Subjects greater than 70 kg were started on 5 mg/day. Dosage was titrated at Visit 3, 5, 6, or 7 based on YGTSS and CGI-TS ratings at the discretion of the investigator. Subjects who showed evidence of response (reduction in CGI-TS by 1-2 points)remained on the same dose. Subjects who did not show evidence of response could be increased: Subjects between 25-50 kg were could be increased 1.25 mg/day at each titration visit, Subjects between 50-70 kg could be increased 2.5 mg/day at each titration visit, and Subjects greater than 70 kg could be increased 5 mg/day at each titration visit.
Period: Overall Study
Arm/Group | Aripiprazole
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Sample: Sample of children and adolescents that enrolled in study to receive active medication. This was not a placebo controlled study.
Arm/Group | Sample
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.36 (3.33)
Gender [Count of Participants; unit: Participants]
  Female | 1
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Calculating Difference Between Means (Baseline and Endpoint Scores on the Yale Global Tic Severity Scale Subscales)
Description: The Yale Global Tic Severity Scale (YGTSS) is a clinical rating instrument that was designed for use in studies of Tourette's syndrome and other tic disorders. The YGTSS provides an evaluation of the number, frequency, intensity, complexity, and interference of motor and phonic symptoms. The maximum YGTSS Global score is 100, while the maximum motor score is 25, the maximum vocal score is 25, and the maximum impairment score is 50. Higher scores indicate more severe tics.
Time Frame: 8 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group 1 - Baseline: Sample of children and adolescents that enrolled in study to receive active medication at baseline.
- Group 1 - Endpoint: Sample of children and adolescents that enrolled in study to receive active medication at endpoint prior to down titration.
Arm/Group | Group 1 - Baseline | Group 1 - Endpoint
Number analyzed (Participants) | 11 | 11
units on a scale
  YGTSS Motor Tic | 15.82 (4.40) | 9.73 (2.76)
  YGTSS Vocal Tic | 12.36 (7.10) | 7.00 (5.76)
  YGTSS Total Tic | 28.18 (7.74) | 16.73 (7.54)
  YGTSS Global Severity | 61.82 (13.49) | 33.73 (15.18)
Statistical Analysis 1: Comparison: Group 1 - Baseline vs Group 1 - Endpoint; Group 1 Baseline vs. Endpoint; Test type: Superiority or Other; p < .05, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = .003 — YGTSS Global Severity score (M=61.8 SD=13.49) declined significantly to end point (M=33.7 SD=15.18; p=0.003)

2. Secondary Outcome: Clinical Global Impression Severity Scores
Description: The Clinical Global Impression scale (CGI) is a classic instrument for making global assessments. This scale yields three different measures: 1. Severity of illness (7-point scale, with 7 being the most impaired; assessment of patient's current symptom severity, referred to here as CGIs), 2. Global improvement (7-point scale, with 7 being the most impaired; comparison of patient's baseline condition with his/her current condition, referred to here as CGIi), 3. Efficacy index (4 point x 4 point rating scale, comparison of patient's baseline condition with a ratio of current therapeutic benefit to severity of side effects)
Time Frame: 24 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 - Baseline | Group 1 - Endpoint
Number analyzed (Participants) | 11 | 11
units on a scale | 4.45 (0.52) | 3.18 (0.60)
Statistical Analysis 1: Comparison: Group 1 - Baseline vs Group 1 - Endpoint; Mean scores baseline to endpoint; Test type: Superiority or Other; p < .05, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = .004 — Mean (SD) CGI-Tic severity scores reduced significantly from (M=4.45 SD=0.52) (moderate-marked) at baseline to (M=3.18 SD =0.60) (mild) at end point ( p=0.004)

ADVERSE EVENTS:
Arm/Group | Sample
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 11/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sample (N=11)
Headache (General disorders) | 11 (34)
Muscle, bone, or joint pain condition (Musculoskeletal and connective tissue disorders) | 10 (31)
Appetite increase/weight gain (General disorders) | 7 (27)
Stomach discomfort (Gastrointestinal disorders) | 9 (26)
Tiredness/fatigue (General disorders) | 8 (23)
Dizziness (General disorders) | 9 (18)
Appetite decrease/weight loss (General disorders) | 6 (12)
Drowsiness/sedation (General disorders) | 7 (13)
Dry mouth (General disorders) | 4 (10)

LIMITATIONS AND CAVEATS:
All subjects failed to respond to previous tic medications so could have unique tic symptoms, small sample size, and this was an open-label study, so we did not have a comparison group nor were we blinded to treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes